CLINICAL TRIAL: NCT07072182
Title: Evaluation of the Effect of Different Biomaterials on Palatal Wound Healing. A Randomized Controlled Clinical Study
Brief Title: Evaluation of the Effect of Different Biomaterials on Palatal Wound Healing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma saad saad mahmoud elsherbini (Other)
Responsible Party: Sponsor-Investigator, Fatma saad saad mahmoud elsherbini, PhD, Lecturer, Oral Medicine, Periodontology, Diagnosis, and Oral Radiology Department,, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M0101025OM
Record Dates: First submitted 2025-07-05; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Heal Wound; VAS Will be Used to Assess Pain Postoperative
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (No Intervention): Palatal wound will be left to heal spontaneously
- study group 1 (Experimental): Palatal wound will be covered with Composite stent
  Interventions: Device: Palatal wound will be covered with Composite stent
- study group 2 (Experimental): Palatal wound will be covered with PRF
  Interventions: Combination Product: Palatal wound will be covered with PRF
- study group 3 (Experimental): Palatal wound will be covered with Ora-aid patch
  Interventions: Device: Palatal wound will be covered with Ora-aid patch

INTERVENTIONS:
Device: Palatal wound will be covered with Ora-aid patch — Palatal wound will be covered with Ora-aid patch
  Other Names: ora aid
  Arms: study group 3
Device: Palatal wound will be covered with Composite stent — Palatal wound will be covered with Composite stent
  Arms: study group 1
Combination Product: Palatal wound will be covered with PRF — Palatal wound will be covered with PRF
  Other Names: prf
  Arms: study group 2

SUMMARY:
All study subjects will sign written informal consent form before enrolment.

They will be divided into four groups, 10 patients each:

* Group I: Palatal wound will be left to heal spontaneously,
* Group II: Palatal wound will be covered with Composite stent,
* Group III: Palatal wound will be covered with PRF,
* Group IV: Palatal wound will be covered with Ora-aid patch. III- Surgical Procedures: -
* After harvesting the palatal soft tissue graft with the standardized dimensions (12 × 7 mm) of the graft for all patients. Graft thickness was standardized as well to be approximately 1.5 to 2 mm and confirmed with a caliper at 3 points (ends and centre of the graft). Fixing of the graft at the recipient site will be performed, back to the donor site for management, the blood clot will be wiped with gauze, then placement of different materials according to each group.
* The dressing will be then pressed gently for 10 seconds, to aid its adherence to the wound. Fixation of the patch will be followed, using 5/0 propylene suture, with performing sling horizontal figure eight suture technique.

ELIGIBILITY:
Inclusion Criteria:-

* Patients who are indicated for soft tissue augmentation procedures, either with root coverage or to increase the deficient keratinized tissue,
* Medically free patients,
* Non-smokers and
* Patients with good oral hygiene. Exclusion Criteria:-
* Pregnant or lactating females,
* Patients with untreated periodontal condition and
* Patients with uncontrolled systemic condition.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Wound healing assessment | From enrollment to the end of treatment at 4 weeks
  The parameters of tissue color, bleeding response to palpation, presence of granulation tissue, characteristics of the incision margins, and the presence of suppuration were evaluated as this index assesses wound healing using scores from 1 to 5: a wound with very poor healing receives a score of 1, whereas excellent healing gets a score of 5.
Pain using the visual analogue scale | From enrollment to the end of treatment at 4 weeks
  Patients were asked about their pain levels, swelling, and other experiences related to the surgical techniques and instruments to assess postoperative pain. The perceived discomfort was rated using a VAS, which is marked at two endpoints: "no discomfort" at one end (score of 0) and "unbearable discomfort" at the other end (score of 10). Patients completed the questionnaires on the 1st, 2nd, 4th, 7th, and 14th days after their surgery

SECONDARY OUTCOMES:
Patient satisfaction through direct communication | From enrollment to the end of treatment at 4 weeks
  Patient satisfaction (PS) was evaluated using a three-point rating scale: 3 for fully satisfied, 2 for satisfied, and 1 for unsatisfied. Each patient was asked about their satisfaction with the following patient-centered criteria: root coverage achieved, relief from dentinal hypersensitivity, color of the gingiva, shape and contour of the gingiva, surgical procedure (including pain during surgery and discomfort related to the duration of the procedure and the operator's handling), post-surgical phase (including pain, swelling, and any postoperative complications), and cost-effectiveness (patients were asked if they felt the treatment justified the time and money spent). This approach aimed to gather comprehensive feedback on the overall patient experience

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university Faculty of dentistry, Al Mansurah, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: No